CLINICAL TRIAL: NCT03216538
Title: A Phase I/II, Single-center, Randomized Double Masked Placebo Controlled Study to Evaluate the Safety and Efficacy of Treatment With AS101 1% Oral Solution in Patients With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Efficacy of AS101 1% Oral Solution in Patients With Neovascular Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Feramda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS101 AMD# 1ֹ
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate; Solutions

STUDY DESIGN:
Intervention Model Description: On day 1 patients will be randomly allocated to one of the two following study arms in a 1:1 ratio and in a masked manner: (1) AS101 1% oral solution (2) Placebo oral solution. Patients of both study arms will be instructed on how to administer orally the drug at home once daily for 24 weeks. Patients will stop taking the study oral solution at week 24 treatment visit.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, caregivers and Investigators will be masked to the nature of the treatment until all patients completed participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AS101 1% oral solution (Active Comparator): Daily dose 0.4 ml administered orally
  Interventions: Drug: AS101 1% oral solution
- Placebo (Placebo Comparator): Daily dose of 0.4 ml administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AS101 1% oral solution — 0.4 ml daily p.o.
  Arms: AS101 1% oral solution
Drug: Placebo — 0.4 ml daily p.o.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AS101 1% oral solution as compared to placebo in patients with neovascular Age-Related Macular Degeneration (AMD).

AMD Patients who underwent 3 consecutive intravitreal anti VEGF injections and have sub retinal or intraretinal fluid at day 1 of study will be treated orally by AS101 1% solution or placebo once daily for 24 weeks and will be tested for sub retinal or intraretinal fluid every 4 weeks by OCT examination. In case of fluid in macula anti intravitreal anti VEGF injections will be given the same day as needed (PRN). Safety evaluation will be assessed by adverse events related to treatment of 1% AS101 oral solution or placebo. Efficacy will be evaluated in terms of duration of fluid free macula in the AS101 treated group as as compared to placebo treated group;

DETAILED DESCRIPTION:
A Phase I/II, single-center, randomized double masked placebo controlled study to evaluate the safety and efficacy of AS101 1% oral solution or placebo once daily for 24 weeks in treating patients with neovascular AMD.

Following confirmation of patient eligibility (as detailed in in the inclusion criteria), patients who meet all of the inclusion and exclusion criteria will be enrolled.

On day 1 patients will be randomly allocated to one of the two following study arms in a 1:1 ratio and in a masked manner: (1) AS101 1% oral solution (2) Placebo oral solution. Patients of both study arms will be instructed on how to administer orally the drug at home once daily for 24 weeks. Patients will stop taking the study oral solution at week 24 treatment visit.

In case of existence of fluid in macula, determined as intra retinal or sub-retinal fluid in the macula (as required in inclusion criteria) the standard to care anti-VEGF intravitreal therapy (Lucentis or Avastin, same as the treatment prior to study start) will be injected by a pro re nata (PRN).

Every 4 weeks the investigator will assess if a patient has a fluid free macula based on clinical evaluation, OCT and FA findings In case of fluid in macula the standard of care anti intravitreal anti VEGF injections (Lucentis or Avastin, same as the treatment prior to study start) will be given the same day by a pro re nata (PRN).

The investigator will monitor the occurrence of any adverse event. The study will be completed at week 24 and the study drug, 1% AS101 oral solution or placebo, will be collected from patients.

At week 28 (4 weeks after treatment completion) all patients will be invited for safety assessment.

If the investigator determines that there is a disease progression study therapy is to be discontinued prior to 24 weeks of treatment. Last observation carried forward (LOCF) technique will be used to analyze such patients.

Efficacy will be evaluated in terms of duration of fluid free macula in the AS101 treated group as compared to placebo treated group;

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with CNV from AMD in one or both eyes and eligible for any anti-VEGF treatment in one or two study eyes.
2. Patient is 50 years of age or older.
3. Patient underwent at least 3 consecutive Intravitreal anti VEGF injections of the same kind , Ranibizumab (Lucentis) or Bevacizumab (Avastin) in the study eye and have sub retinal or intraretinal fluid at day 1, as found in OCT examination.
4. Patient must understand and sign the IRB-approved informed consent document for the study.
5. Patient must have BCVA of at least 20/200 in the study eye.
6. While unlikely, female patients of childbearing potential must not be pregnant or breast-feeding an must be willing to undergo serum pregnancy tests throughout the study. Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child-bearing potential.
7. Both female patients of childbearing potential and male patients able to father a child must have (or have a partner who has) an acceptable method of contraception (such as hormonal or condoms) throughout the course of the study and for 4 weeks after the last study medication administration.
8. Patient must be willing and able to comply with the study procedures.

Exclusion Criteria:

1. Patient exhibits evidence of retinal angiomatous proliferation in the study eye.
2. Patient has retinal-choroidal anastomosis in the study eye.
3. Patient has a history of treatment for CNV in the study eye with verteporfin, transpupillary thermotherapy, laser photocoagulation, external beam radiation therapy, or other local treatment (such as submacular surgery).
4. Patient has a history of systemic, periocular or intraocular steroid use at any time during the 12 weeks prior to enrollment.
5. Patient has a corneal melting, necrotizing keratitis/scleritis, scleritis of an infectious etiology or impending vision loss.
6. Patient has a known underlying systemic disease with evidence of a serious or potentially lethal uncontrolled active disease in one or more extraocular organ systems for which a defined effective medical regimen is indicated.
7. Patient has active pulmonary tuberculosis or active viral hepatitis.
8. Patient has a significant active infection.
9. Patient has significant renal or hepatic function impairment greater than mild (grade 2) as per CTCAE v4.0 or hypercholesterolemia uncontrolled by medication and/or diet.
10. Pregnant patients or lactating.
11. Patient has a history of malignancy within the past two years other than non-melanoma skin cancer.
12. Patient has an autoimmune systemic disease requiring immunosuppressive treatment or patient has other medical condition that renders the patient immunocompromised.
13. Patient received a live vaccine within past six weeks.
14. Patient has significant ocular or periocular inflammation or infection in either eye.
15. Patient has the presence of active or inactive toxoplasmosis in the study eye.
16. Patient is scheduled for surgery during study.

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence and severity of treatment emerged ocular and non-ocular adverse events | 28 weeks
  as assessed by visual acuity measurement, ophthalmic examinations, vital signs, laboratory tests and adverse events related to 1% AS101 oral solution as compared to placebo.

SECONDARY OUTCOMES:
Duration of fluid free macula in average | 28 weeks
  As assessed every 4 weeks by OTC
Duration of fluid free macula | 24 weeks
  Proportion in number of patients that had an increase in the duration of fluid free macula;
Best corrected visual acuity (BCVA) | 24 Weeks
  changes in BCVA using the Early treatment diabetic retinopathy study (ETDRS) chart;
Central retinal subfield thickness (CRT) | 24 weeks
  CRT as measured by optical coherence tomography (OCT);
Lesion size in the macula | 24 weeks
  Changes as demonstrated by fluorescein angiography (FA) if feasible;

CONTACTS AND LOCATIONS:
Locations (1):
- Meir MC, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No